CLINICAL TRIAL: NCT03028727
Title: Diode Laser Therapy As An Adjunct To Non-Surgical Management Of Chronic Periodontitis - A Pilot Study
Brief Title: Diode Laser Therapy As An Adjunct To Scaling And Root Planing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KLE Society's Institute of Dental Sciences (Other)
Responsible Party: Principal Investigator, Veena H.R, Reader, Department of Periodontics, KLE Society's Institute of Dental Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KLESocietyIDS
Record Dates: First submitted 2017-01-07; First posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Root Planing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ultrasonic Scaling, Root planing (Active Comparator): Ultrasonic Scaling and Root planing at day 0 and at 1 week.
  Interventions: Procedure: Ultrasonic Scaling and root planing
- 980 nm diode Laser irradiation (Experimental): Irradiation of periodontal pockets with with 980 nm diode Laser after scaling and root planing at day 0 and after 1 week.
  Interventions: Procedure: Ultrasonic Scaling and root planing; Procedure: 980 nm diode laser irradiation

INTERVENTIONS:
Procedure: Ultrasonic Scaling and root planing — Procedure of scaling and root planing at day 0 and at 1 week
Procedure: 980 nm diode laser irradiation — Procedure of scaling and root planing and application of 980 nm diode laser at day 0 and at 1 week
  Arms: 980 nm diode Laser irradiation

SUMMARY:
Laser therapy has been proposed as a novel treatment option in controlling subgingival microorganisms. This randomized controlled clinical trial evaluates the effect of 980nm diode laser as an adjunct to scaling and root planing (SRP) in the management of chronic periodontitis (CP).

DETAILED DESCRIPTION:
Conventional mechanical debridement can achieve a temporary decrease in the subgingival levels of Pg along with other pathogens. However, mechanical therapy alone may fail to eliminate pathogenic bacterial niches in inaccessible areas like deep pockets, root concavities, furcation areas etc. In search of more efficient and less traumatic techniques to improve periodontal healing, researchers proposed the use of lasers in periodontal therapy.

The adjunctive use of lasers with conventional tools may facilitate treatment and have the potential to improve healing. The diode laser is highly absorbed in hemoglobin and other pigments and is excellent for use in soft tissue surgical procedures.Laser application in improving clinical outcome in periodontal therapy, needs to be further investigated with well designed clinical trials. The investigators attempted to evaluate the efficacy of diode laser as an adjunct to SRP in the management of CP by evaluating clinical parameters coupled with quantitative estimation of P.gingivalis using Real-time Polymerase chain reaction (RT-PCR) assay.

ELIGIBILITY:
Inclusion Criteria:

* 40 systemically healthy subjects diagnosed with generalized moderate CP in the age group of 30 to 50 years.
* Minimum of 20 teeth having atleast two non-adjacent sites per quadrant with probing pocket depth of ≥ 5mm and clinical attachment loss of 3- 4 mm

Exclusion Criteria:

* Patients who had undergone periodontal therapy 6 months prior to the commencement of the study.
* Subjects on antibiotics or immunosuppressants.
* Chronic smokers, alcoholics, smokeless tobacco users.
* Subjects with acute illnesses/acute intraoral lesions.
* Pregnant women
* Subjects who had undergone extensive restorative dental treatment.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change in levels of P.gingivalis | 14 weeks
  Microbial profile was assessed using PCR at baseline, 4-6 weeks and 12-14 weeks post treatment in both the study groups.

SECONDARY OUTCOMES:
Change in gingival index | 14 weeks
  Gingival index by Loe and Silness was assessed at baseline, 4-6 weeks and 12-14 weeks post treatment in both the groups
Change in plaque index | 14 weeks
  Plaque index by Silness and Loe was assessed at baseline, 4-6 weeks and 12-14 weeks
Change in probing pocket depth | 14 weeks
  Probing pocket depth was assessed at baseline, 4-6 weeks and 12-14 weeks
Change in clinical attachment level | 14 weeks
  Clinical attachment level was assessed at baseline, 4-6 weeks and 12-14 weeks

IPD SHARING:
Plan to Share IPD: No